CLINICAL TRIAL: NCT00860158
Title: A Phase II Study of Neoadjuvant Dasatinib Plus LHRH Analogue Therapy in High-Risk Localized Prostate Cancer
Brief Title: Neoadjuvant Dasatinib Plus LHRH Analogue Therapy in High-Risk Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual; closed by funder
Sponsor: Noah Hahn, M.D. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Noah Hahn, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GU07-124
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib; Leuprolide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Assignment (Experimental): Neoadjuvant dasatinib plus leuprolide acetate followed by radical prostatectomy
  Interventions: Drug: Dasatinib; Drug: Leuprolide Acetate (LHRH Analogue); Procedure: Radical Prostatectomy

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 100 mg administered once daily per oral route for 28 consecutive days
Drug: Leuprolide Acetate (LHRH Analogue) — Leuprolide acetate 7.5 mg administered subcutaneously on day 1 every 28 days (+ 7 days).
Procedure: Radical Prostatectomy — Radical prostatectomy should be performed no sooner than 8 hours but preferably within 24 hours of the last administered dasatinib dose.

SUMMARY:
This trial will investigate the activity of dasatinib plus LHRH analogue therapy in high-risk localized prostate cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Dasatinib -100 mg administered once daily per oral route for 28 consecutive days.
* Leuprolide acetate - 7.5 mg administered subcutaneously on day 1 every 28 days (+ 7 days).

The 28 days of dasatinib and leuprolide injection (plus the time required to recover from toxicity if encountered) is defined as a cycle. Patients will be treated for up to a maximum of 3 cycles of dasatinib and leuprolide acetate.

Radical Prostatectomy should be performed no sooner than 8 hours but preferably within 24 hours of the last administered dasatinib dose. All attempts should be made for the patient to have their surgery after 8 hours but within 24 hours of their last dose of dasatinib. If surgery delay is imperative, dasatinib therapy should continue until at least 24 hours before planned surgery.

Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Hematopoietic:

* Hemoglobin (Hgb) ≥ 8.0 g/dL
* Platelets ≥ 100 K/mm3
* Absolute neutrophil count (ANC) ≥ 1.0 K/mm3

Hepatic:

* Total bilirubin < 2.0 X Upper Limit Normal (ULN)
* Aspartate aminotransferase (AST) < 2.5 X ULN
* Alanine aminotransferase (ALT) < 2.5 X ULN

Renal:

* Calculated creatinine clearance of ≥ 60 cc/min using the Cockcroft-Gault formula

Cardiovascular:

* No uncontrolled angina, congestive heart failure or myocardial infarction within 6 months prior to registration for protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Clinical stage T1-T3a disease.
* Must be willing to have a tumor biopsy, if previous tumor tissue unavailable for tumor marker analysis.
* Kattan pre-operative nomogram-predicted (based on stage, Prostate Specific Antigen (PSA) and Gleason score) 5-year risk of recurrence-free survival of 80% or less
* Must be deemed eligible for radical prostatectomy.
* Must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.

Exclusion Criteria:

* No evidence of regional, lymph node or distant metastasis on clinical or radiological assessments. All baseline radiology studies must be performed within 28 days prior to registration for protocol therapy.
* No prior malignancy in the past 2 years except for basal cell and squamous cell carcinoma of the skin. Other cancers with low potential for metastasis, such as in situ cancers (e.g., Grade 1, TA TCC (low grade superficial bladder cancer), and colonic polyp with focus of adenocarcinoma) can be enrolled after approval from the Sponsor Investigator.
* No prior hormonal therapy with the exception of oral 5-alpha-reductase inhibitors (finasteride, dutasteride, etc.). Patients who have received prior oral anti-androgen therapies (bicalutamide, flutamide, nilutamide, etc.), prior LHRH agonist therapy (leuprolide, goserelin acetate, etc.), or prior orchiectomy are ineligible.
* No prior systemic chemotherapy or radiotherapy for prostate cancer is allowed. Transurethral resection of the prostate for benign prostatic hypertrophy (BPH) and oral alpha-blockers (terazosin, tamsulosin, doxazosin) are permitted.
* No history of hemorrhage or thrombotic events (cerebrovascular accident, deep vein thrombosis, pulmonary embolism, etc.) within 6 months prior to registration for protocol therapy.
* No history of diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
* No history of diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) of registration on protocol therapy.
* No history of ongoing or recent (≤ 3 months of registration on protocol therapy) significant gastrointestinal bleeding
* No ongoing anti-coagulation and/or anti-platelet therapies allowed.
* No unresolved pleural or pericardial effusion of any grade within 3 months of registration for protocol therapy.
* No uncontrolled angina, congestive heart failure or MI within 6 months prior to registration for protocol therapy.
* No diagnosed congenital long QT syndrome.
* No history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes).
* No prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* Following medications must be discontinued at least 7 days prior to registration for protocol therapy and be withheld for the duration of dasatinib therapy:
* Drugs that are generally accepted to have a risk of causing Torsades de Pointes
* Patient must not be receiving any prohibited CYP3A4 inhibitors /inducers/ substrates
* Anti-coagulation and/or anti-platelet therapies - to avoid potential bleeding risks.
* No major surgical procedure, open biopsy, or significant trauma within 28 days prior to registration for protocol therapy.
* Ability to comply with study and/or follow-up procedures and requirements.
* No treatment with any investigational agent for any medical condition within 28 days prior to registration for protocol therapy.
* No clinically significant infections or any other condition which, in the investigator's opinion, deems the patient an unsuitable candidate to receive the study drug.
* Ability to take oral medication (dasatinib must be swallowed whole).
* No known history of hypokalemia that cannot be corrected prior to registration on protocol therapy.
* No known history of hypomagnesemia that cannot be corrected prior to registration on protocol therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Hahn, M.D., Study Chair — Hoosier Cancer Research Network
Locations (6):
- United States (6):
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Neoadjuvant dasatinib plus leuprolide acetate followed by radical prostatectomy
  Dasatinib: Dasatinib 100 mg administered once daily per oral route for 28 consecutive days
  Leuprolide Acetate (LHRH Analogue): Leuprolide acetate 7.5 mg administered subcutaneously on day 1 every 28 days (+ 7 days).
  Radical Prostatectomy: Radical prostatectomy should be performed no sooner than 8 hours but preferably within 24 hours of the last administered dasatinib dose.
Period: Overall Study
Arm/Group | Experimental Arm
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: To Estimate the Pathologic Complete Response (pCR) Rate
Time Frame: 18 months
Population: No participants were analyzed for pCR due to study termination
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

2. Secondary Outcome: To Estimate Partial Pathologic Responses (pPR)
Time Frame: 18 months
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

3. Secondary Outcome: To Estimate PSA Response Rate
Time Frame: 18 months
Population: Data for this secondary objective was not collected or analyzed.
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

4. Secondary Outcome: To Estimate Progression Free Survival
Time Frame: 18 months
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

5. Secondary Outcome: To Evaluate the Impact of Dasatinib Plus LHRH on Expression of Selected Biomarkers
Time Frame: 18 months
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

6. Secondary Outcome: To Estimate Safety and Tolerability of LHRH Plus Dasatinib
Time Frame: 18 months
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm Assignment
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Assignment (N=1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated due to slow accrual and no results were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No